CLINICAL TRIAL: NCT01111461
Title: An Open-Label, Single-Arm, Multicenter Phase II Study of E7080 (Lenvatinib) in Subjects With Advanced Endometrial Cancer and Disease Progression Following First-Line Chemotherapy
Brief Title: Study of Lenvatinib in Subjects With Advanced Endometrial Cancer and Disease Progression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7080-G000-204
Record Dates: First submitted 2010-04-16; First posted 2010-04-27 (Estimated); Results first posted 2016-04-18 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2016-11

CONDITIONS: Endometrial Cancer
Keywords: Advanced Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenvatinib 24 mg (Experimental): Participants with advanced endometrial cancer and disease progression following platinum-based, first line chemotherapy.
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib 24 mg administered orally, once daily continuously in 28-day cycles to participants with advanced endometrial cancer and disease progression following first-line chemotherapy. Participants continued to receive study drug until disease progression, development of unacceptable toxicity or withdrawal of consent. 'Treatment interruption and subsequent dose reduction' was allowed for participants who experienced lenvatinib-related toxicity.
  Other Names: E7080, Lenvima

SUMMARY:
To assess the objective response rate (ORR: complete response + partial response [CR+ PR]) of E7080 in subjects with unresectable endometrial cancer and disease progression following platinum-based, first-line chemotherapy. .

ELIGIBILITY:
Inclusion criteria:

1. Histologically confirmed diagnosis of endometrial carcinoma.
2. Radiographic evidence of disease progression according to modified RECIST 1.1 after 1 prior systemic, platinum-based chemotherapy regimen for recurrent metastatic or primary unresectable endometrial carcinoma for which no surgical or radiotherapy treatment option exists.
3. Measureable disease meeting the following criteria:

   * At least 1 lesion of greater than 1.0 cm in the longest diameter for a non-lymph node or greater than 1.5 cm in the short-axis diameter for a lymph node which is serially measureable according to modified RECIST 1.1 using computerized tomography / magnetic resonance imaging.
   * Lesions that have had external beam radiotherapy (EBRT) or loco-regional therapies such as radiofrequency ablation must show evidence of progressive disease based on modified RECIST 1.1 to be deemed a target lesion.
4. Eastern Cooperative Oncology Group (ECOG) performance status less than 2.
5. Adequate controlled blood pressure (BP) with or without antihypertensive medications, defined as BP less than 150/90 mmHg at screening and no change in antihypertensive medications within 1 week prior to the Screening Visit.
6. Adequate renal function defined as calculated creatinine clearance greater than 30 mL/min per the Cockcroft and Gault formula.
7. Adequate bone marrow, blood coagulation, and liver functions, as defined in the study protocol.
8. Negative serum or urine pregnancy test for women of reproductive potential.

Exclusion criteria:

1. Brain or leptomeningeal metastases, including stable metastases.
2. More than 1 prior systemic chemotherapy regimen for recurrent metastatic or primary unresectable endometrial carcinoma or any treatment targeting vascular endothelial growth factor (VEGF)-directed angiogenesis. No restriction regarding prior adjuvant chemotherapy or hormonal therapy.
3. Prior systemic anti-tumor therapy within 3 weeks.
4. Not fully recovered from prior radiotherapy based on investigator judgement.
5. Participants with greater than 1+ proteinuria on urine dipstick testing to undergo 24-hour urine collection for quantitative assessment of proteinuria. Participants with greater than 1 gm will be ineligible.
6. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association Class II; unstable angina; myocardial infarction or stroke within 6 months of the first dose of study drug; cardiac arrhythmia requiring medical treatment.
7. Prolongation of QTc interval greater than 480 msec.
8. Bleeding disorder or thrombotic disorders requiring anticoagulant therapy, such as warfarin, or similar agents requiring therapeutic INR monitoring (treatment with low molecular weight heparin [LMWH] allowed).
9. Active hemoptysis within 3 weeks prior to the first dose of study drug.
10. Females who are pregnant or breast feeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2010-03; Primary Completion 2012-05 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eisai Medical Services, Study Director — Eisai Limited
Locations (78):
- United States (36):
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Los Angeles, California
  - Honolulu, Hawaii
  - Arlington Heights, Illinois
  - Niles, Illinois
  - Boston, Massachusetts
  - Detroit, Michigan
  - Burnsville, Minnesota
  - Edina, Minnesota
  - Maplewood, Minnesota
  - Minneapolis, Minnesota
  - Saint Paul, Minnesota
  - Woodbury, Minnesota
  - St Louis, Missouri
  - Morristown, New Jersey
  - New York, New York
  - Chapel Hill, North Carolina
  - Cleveland, North Carolina
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Eugene, Oregon
  - Portland, Oregon
  - Springfield, Oregon
  - Tualatin, Oregon
  - Charleston, South Carolina
  - Austin, Texas
  - Bedford, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Tyler, Texas
  - Newport News, Virginia
  - Norfolk, Virginia
  - Virginia Beach, Virginia
  - Vancouver, Washington
- Belgium (11):
  - Arlon
  - Charleroi
  - Duffel
  - Ghent
  - Kortrijk
  - Leuven
  - Liège
  - Namur
  - Ostend
  - Roeselare
  - Yvoir
- Bulgaria (5):
  - Pleven
  - Plovdiv
  - Sofia
  - Varna
  - Veliko Tarnovo
- Hungary (2):
  - Budapest
  - Győr
- Poland (3):
  - Lublin
  - Poznan
  - Warsaw
- Romania (4):
  - Brasov County
  - Bucharest
  - Cluj County
  - Dolj County
- Russia (12):
  - Kazan'
  - Nizhny Novgorod
  - Orenburg
  - Pyatigorsk
  - Saint Petersburg
  - Sochi
  - Stavropol
  - Syktyvkar
  - Tomsk
  - Tula
  - Ufa
  - Vladivostok
- Ukraine (5):
  - Chernihiv
  - Donetsk
  - Kharkiv
  - Kyiv
  - Zaporizhia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 167 participants were screened for entry into the study. Of these 167 participants, 133 participants met inclusion/exclusion criteria and were treated with at least 1 dose of lenvatinib 24 mg.
Groups:
- Lenvatinib 24 mg: Lenvatinib hard capsules, 24 mg (two 10-mg capsules and one 4-mg capsule) were self-administered orally once a day in the morning (without regard to food intake) in 28-day cycles. Dose reduction or interruption was allowed for participants who experienced lenvatinib-related toxicity.
Period: Overall Study
Arm/Group | Lenvatinib 24 mg
Started | 133
Completed | 82 (On treatment at data cut-off or on treatment until disease progression)
Not Completed | 51
Not completed — Adverse Event | 32
Not completed — Participant choice | 11
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1
Not completed — Other | 6

BASELINE CHARACTERISTICS:
Groups:
- Lenvatinib 24 mg: Lenvatinib 24 mg was administered orally, once daily continuously in 28-day cycles
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133
  Male | 0
Prior Platinum-based Chemotherapy Regimen [Number; unit: Participants] — Participants could have received more than one prior platinum based chemotherapy regimen.
  Participants
    Carboplatin | 80
    Cisplatin | 47
    Cisplatin w/Doxorubicin | 4
    Taxol [Paclitaxel] w/Carboplatin | 10

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR) based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 for target lesions assessed by magnetic resonance imaging/computed tomography (MRI/CT) scans, as determined by independent radiologic review. BOR of CR was confirmed by a subsequent CR assessment at least 4 weeks later. BOR of PR was confirmed by a subsequent CR or PR assessment at least 4 weeks later. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (target or non-target) had to be reduced in short axis to <10 mm. PR was defined as at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum of diameters. The null hypothesis ORR was ≤10% was tested using 1-sided exact test of a single proportion, at 1-sided 0.05 level. ORR was presented with corresponding 2-sided, 95% confidence interval (CI). ORR=CR+PR
Time Frame: From the date of first administration of study treatment until all participants completed a minimum of 6 cycles (28-day cycles) or discontinued treatment prior to the end of Cycle 6 (as of 21 May 2012 data cut-off)
Population: Full Analysis Set (Intent-to-Treat [ITT] Analysis Set) was used and included all participants who received at least 1 dose lenvatinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 133
Percentage of participants | 14.3 [8.8 to 21.4]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was measured as the time from the date of first administration of study treatment until the date of first documentation of disease progression or date of death (whichever occurred first), as determined by independent radiologic review (IRR) and Investigator based on RECIST 1.1. Disease progression per RECIST v1.1 was defined as at least a 20% relative increase and 5 mm absolute increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) recorded since the treatment started or the appearance of 1 or more new lesions.
Time Frame: From date of first administration of study treatment until the date of first documentation of disease progression or date of death, if death occurred prior to disease progression or up to approximately 26 months (as of 21 May 2012 data cut-off)
Population: Full Analysis Set (ITT Population) included all participants who received at least 1 dose of lenvatinib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 133
Months
  Determined by IRR | 5.6 [3.7 to 6.3]
  Determined by Investigator | 5.4 [3.7 to 6.7]

3. Secondary Outcome: Overall Survival (OS)
Description: OS was the length time in months from the date of first treatment until the date of death from any cause. If death was not observed, OS was censored at the last known alive date or data cut-off. Additional survival follow-up data was collected for all participants who had not withdrawn consent and were alive at the time of the initial survival follow-up as of 26 Nov 2012 data cut-off. Participants who were lost to follow-up at the time of the initial assessment may have been contacted again at the investigator's discretion. Updated survival (based on 26 Nov 2012 cut-off) was derived for these participants if the contact was made successfully.
Time Frame: From date of first administration of study treatment until the date of death, or up to approximately 32 months (as of 26 Nov 2012 data cut-off)
Population: Full Analysis Set (ITT Population) included all participants who received at least 1 dose of lenvatinib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 133
Months | 10.6 [8.9 to 14.9]

4. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants with BOR of CR or PR or stable disease (SD) based on RECIST 1.1 and SD lasting greater than or equal to 7 weeks, as determined by IRR and Investigator.
Time Frame: From date of first administration of study treatment until the date of first documentation of disease progression or date of death, if death occurred prior to disease progression, or up to approximately 26 months (as of 21 May 2012 data cut-off)
Population: Full Analysis Set (ITT Population) included all participants who received at least 1 dose of lenvatinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 133
Percentage of participants
  Determined by IRR | 60.9 [52.1 to 69.2]
  Determined by Investigator | 66.2 [57.5 to 74.1]

5. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR was defined as the percentage of participants with BOR of CR or PR or durable stable disease (dSD) [CR + PR + dSD] based on RECIST 1.1. The dSD rate was defined as the percentage of participants with dSD (based on RECIST 1.1 and defined as SD lasting greater than or equal to 23 weeks), as determined by the IRR and Investigator.
Time Frame: as for outcome 4
Population: Full Analysis Set (ITT Population) included all participants who received at least 1 dose of lenvatinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 133
Percentage of participants
  Determined by IRR | 37.6 [29.3 to 46.4]
  Determined by Investigator | 44.4 [35.8 to 53.2]

6. Secondary Outcome: Number of Participants With Adverse Events (AEs) /Serious Adverse Events (SAEs) as a Measure of Safety and Tolerability of Lenvatinib Tolerability of Lenvatinib
Description: Safety was assessed by monitoring and recording all AEs and SAEs, regular monitoring of hematology, clinical chemistry, and urine values, regular measurement of vital signs, electrocardiograms (ECGs), and echocardiograms.
Time Frame: From the administration of first dose up to 30 days after the last dose, or up to data cut-off (21 May 2012), or up to approximately 26 months.
Population: Safety Analysis Set included all participants who received at least 1 dose of lenvatinib and had at least 1 postbaseline safety evaluation. This was the analysis set for all safety evaluations.
Measure: Number; unit: Participants
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 133
Participants
  AEs | 126
  SAEs | 62

7. Other Pre Specified Outcome: Summary of Plasma Concentration of Lenvatinib
Description: A total of 6 blood samples for pharmacokinetic (PK) analysis were collected from each participant who received lenvatinib once daily.
Time Frame: Predose and 2 hours postdose on Cycle 1 Day 1, Cycle 1 Day 8, and Cycle 2 Day 1
Population: PK analysis set was used and included all participants with an evaluable plasma concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 133
ng/mL
  Cycle 1, Day 1 (Pre-dose) n=132 | 0 (0)
  Cycle 1, Day 1 (2-hour Post-dose) n=132 | 318.9 (242.16)
  Cycle 1, Day 8 (Pre-dose) n=122 | 105.6 (121.66)
  Cycle 1, Day 8 (2-hour Post-dose) n=123 | 352.6 (243.88)
  Cycle 2, Day 1 (Pre-dose) n=107 | 88.63 (78.768)
  Cycle 2, Day 1 (2-hour Post-dose) n=102 | 336.8 (222.56)

8. Other Pre Specified Outcome: Percentage Change From Baseline for the Imaging Biomarker Parameter of the Area Under the Plasma Concentration Curve Blood Normalized (90) (AUCBN (90)) Median for Total Volume
Description: The antiangiogenic and direct antitumor effects of lenvatinib were assessed by analyses of 2 dynamic contrast-enhanced magnetic resonance imaging/diffusion-weighted magnetic resonance imaging (DCE-MRI/DWI MRI) scans obtained on evaluable participants at Baseline and Cycle 1 Day 5. The scans were obtained using standardized acquisition across sites. DWI sequences totaling approximately 30 seconds were acquired during the DCE-MRI scans. Centralized analysis metrics for DCE-MRI included percentage change in initial area under the gadolinium contrast agent time-concentration curve (first 90 seconds, blood normalized) from baseline.
Time Frame: Cycle 1 Day 5
Population: Imaging biomarker analysis set included those participants who received at least 1 dose of lenvatinib and had, at minimum, a baseline and 1 postbaseline evaluable imaging assessment. n = 4 participants with evaluable data.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 4
Percentage change | -34.0 (18.98)

9. Other Pre Specified Outcome: Percentage Change From Baseline in the Contrast Volume Transfer Coefficient (Ktrans) Median
Description: The antiangiogenic and direct antitumor effects of lenvatinib were assessed by analyses of two DCE-MRI/DWI MRI scans obtained on evaluable participants at Baseline and Cycle 1 Day 5. The scans were obtained using standardized acquisition across sites. DWI sequences totaling approximately 30 seconds were acquired during the DCE-MRI scans. Centralized analysis metrics for DCE-MRI included the percentage change in Ktrans for gadolinium chelate movement from the vasculature into the tissue extracellular space from baseline.
Time Frame: Cycle 1 Day 5
Population: Imaging biomarker analysis set included those participants who received at least 1 dose of lenvatinib and had, at a minimum, a baseline and 1 postbaseline evaluable imaging assessment. n = 4 participants with evaluable data.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 4
Percentage change | -41.5 (22.02)

10. Other Pre Specified Outcome: Percentage Change From Baseline in the Apparent Diffusion Coefficient (ADC) Median
Description: The antiangiogenic and direct antitumor effects of lenvatinib were assessed by analyses of two DCE-MRI/DWI MRI scans obtained on evaluable participants at Baseline and Cycle 1 Day 5. The scans were obtained using standardized acquisition across sites. DWI sequences totaling approximately 30 seconds were acquired during the DCE-MRI scans. Centralized analysis metrics for DCE-MRI included the percentage change in ADC for gadolinium chelate movement from the vasculature into the tissue extracellular space from baseline.
Time Frame: Cycle 1 Day 5
Population: Imaging biomarker analysis set included those participants who received at least 1 dose of lenvatinib and had, at a minimum, a baseline and 1 postbaseline evaluable imaging assessment. n = 2 participants with evaluable data.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Lenvatinib 24 mg
Number analyzed (Participants) | 2
Percentage change | 2.1 (2.27)

ADVERSE EVENTS:
Time Frame: From date of administration of first dose up to 30 days after the last dose, or up to data cut-off (21 May 2012), or up to approximately 26 months.
Description: Treatment-emergent adverse events (TEAEs) and serious TEAEs were collected and reported. Safety analysis set included all participants who received at least one dose of study drug. AEs were graded using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Arm/Group | Lenvatinib 24 mg
Serious Adverse Events (participants affected / at risk) | 62/133
Other Adverse Events (participants affected / at risk) | 125/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib 24 mg (N=133)
Abdominal pain (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 3
Colitis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Intestinal obstruction (Gastrointestinal disorders) | 2
Small intestinal obstruction (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Gastrointestinal fistula (Gastrointestinal disorders) | 1
Ileitis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Rectal perforation (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 6
General physical health deterioration (General disorders) | 3
Device leakage (General disorders) | 1
Impaired healing (General disorders) | 1
Multi-organ failure (General disorders) | 1
Pyrexia (General disorders) | 1
Hypertension (Vascular disorders) | 6
Hypotension (Vascular disorders) | 4
Deep vein thrombosis (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Metabolic disorder (Metabolism and nutrition disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Renal failure acute (Renal and urinary disorders) | 6
Azotaemia (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal disorder (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1
Urinary tract infection (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 1
Peridiverticular abscess (Infections and infestations) | 1
Proctitis infectious (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cardiopulmonary failure (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 1
Ejection fraction decreased (Investigations) | 1
Female genital tract fistula (Reproductive system and breast disorders) | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Deafness (Ear and labyrinth disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib 24 mg (N=133)
Anaemia (Blood and lymphatic system disorders) | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 11
Hypothyroidism (Endocrine disorders) | 23
Vision blurred (Eye disorders) | 7
Abdominal distension (Gastrointestinal disorders) | 9
Abdominal pain (Gastrointestinal disorders) | 33
Abdominal pain upper (Gastrointestinal disorders) | 17
Constipation (Gastrointestinal disorders) | 25
Diarrhoea (Gastrointestinal disorders) | 46
Dry mouth (Gastrointestinal disorders) | 15
Dyspepsia (Gastrointestinal disorders) | 7
Flatulence (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 41
Stomatitis (Gastrointestinal disorders) | 30
Vomiting (Gastrointestinal disorders) | 32
Asthenia (General disorders) | 30
Fatigue (General disorders) | 55
Oedema peripheral (General disorders) | 20
Urinary tract infection (Infections and infestations) | 17
Blood thyroid stimulating hormone increased (Investigations) | 8
Weight decreased (Investigations) | 27
Decreased appetite (Metabolism and nutrition disorders) | 45
Dehydration (Metabolism and nutrition disorders) | 8
Hypokalaemia (Metabolism and nutrition disorders) | 17
Hypomagnesaemia (Metabolism and nutrition disorders) | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Dizziness (Nervous system disorders) | 20
Dysgeusia (Nervous system disorders) | 16
Headache (Nervous system disorders) | 35
Insomnia (Psychiatric disorders) | 7
Dysuria (Renal and urinary disorders) | 9
Proteinuria (Renal and urinary disorders) | 28
Vaginal haemorrhage (Reproductive system and breast disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 19
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 27
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13
Alopecia (Skin and subcutaneous tissue disorders) | 7
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 10
Rash (Skin and subcutaneous tissue disorders) | 9
Hypertension (Vascular disorders) | 71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other